CLINICAL TRIAL: NCT05057520
Title: Establish an Evaluation Scale for the Quality of Primary Care in Multi-professional Health Centres and Homes Integrating the Point of View of Patients in Complex Care Situations and Their Caregivers.
Acronym: Qualsoprim_3
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0009
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Patients in Complex Situations
Keywords: Multimorbidity; Exercise coordinated groups (GECO); Caregivers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Completion of the questionnaire by the patient after consultation with the general practitioner

SUMMARY:
The prevalence of multimorbid patients and complex care is increasing in France and elsewhere in the world. It concerns 60% of the over 65 years old. Comprehensive care, the involvement of the patient and his caregivers appear as the solutions for the management of these new care situations. The structures of multi-professional grouping, developing a coordinated exercise (GECO), appear as the privileged place to take care of these patients. These structures become the main place of exercise in France (improved working conditions for professionals, financial incentives, public policy, etc.); they have shown their ability to formulate patient care protocols, to produce coordinated exercise, to better involve the patient and caregivers in their care. The question of improving the quality of care arises. To date, there is no data on the subject apart from some evaluations mainly medico-economic. The patient's place in the evaluation showed his interest with the existence of a proven correlation between patient satisfaction in particular and his compliance and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, followed in primary care centers, able to participate, speaking and understanding French,
* Patient in a complex care situation, benefiting from a multi-professional management (at least two different professionals from the center including the general practitioner),
* No opposition from the patient.

Exclusion Criteria:

* Patient not in a complex care situation
* Patient followed only by the the exercise coordinated group general practitioner
* Refusal to participate
* Patients who have already participated in phase 2 of the Qualsoprim project
* Adults under legal protection or unable to express their consent
* Persons deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed in the primary care center and being in a complex care situation, benefiting from a multi-professional care
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Reliability of questionnaire | 1 day
  The main objective of this phase of the protocol is to confirm on an independent sample the reliability of the primary care quality assessment questionnaire scales provided within the coordinated exercise groups from the point of view of patients in complex care situations, their caregivers and health professionals.

SECONDARY OUTCOMES:
Concurrent validity of questionnaire | 1 day
  Test the concurrent validity by comparison with EUROPEP questionnaire to verify that it does indeed measure the latent trait it is supposed to measure. The EUROPEP questionnaire is a 23-item validated and internationally standardized measure of patient evaluations of general practice care.
Anchor variables | 1 day
  Test anchor variables that can be used later to assess sensitivity to change (comparison of means test if the candidate variable is qualitative and Spearman correlation if it is quantitative).
Standardized scoring guide | 1 day
  To construct a standardized scoring guide if a satisfactory questionnaire is obtained.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Maison de santé de Bannalec, Bannalec
  - Maison de santé de Châteauneuf-du-Faou, Châteauneuf-du-Faou
  - Maison de santé de Coray, Coray
  - Pôle de santé de Lanmeur, Lanmeur
  - Maison de santé de Trébeurden, Trébeurden

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of BrestUH. Requestors will be required to sign and complete a data access agreement.